CLINICAL TRIAL: NCT03309293
Title: Construction and External Validation of a Predictive Clinico-biological Score of the Risk of Venous Thrombosis in Women Under Combined Oral Contraceptives
Acronym: PILGRIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-22; 2017-A01591-52 (Registry Identifier: n°IDRCB)
Record Dates: First submitted 2017-10-05; First posted 2017-10-13 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- controls (Other): biological samples bank
  Interventions: Biological: blood samples
- cases (Experimental)
  Interventions: Biological: blood samples

INTERVENTIONS:
Biological: blood samples — blood samples

SUMMARY:
the investigators hypothesize that some of these polymorphisms contribute to VTE risk in women using COC, and that their screening could to help assess individual risk of VTE before COC prescription.

In order to test this hypothesis the investigators propose to build a predictive score for VTE in women using COC based on clinical and biological factors. To this end the investigators have a large case study (including 766 patients) recruited at the "Centre d'Exploration des Pathologies Hémorragiques et Thrombotiques" (CEHT) of the laboratory of Hematology (La Timone Hospital, Marseille) between 2003 and 2013. The cases had a personal history of documented VTE while using COC (PILGRIM study). A great number of clinical and biological relevant phenotypes in the field of VTE have already been collected (including 14 polymorphisms selected on the basis of their biological plausibility and the existence association studies).To our knowledge it is the largest study specifically conducted in order to assess genetic factors associated with VTE in women using COC. These 766 cases will be compared to 766 controls from the general population (cohort Nutrinet-Santé). Then, the predictive values of the score will be assessed in an independent multicentric validation study that the investigators will set up in the field of this project. Our study should allow a better understanding of the genetic and environmental factors involved in VTE related to COC use. Besides, this project aims to respond to a major public health issue giving an effective tool for the decision of prescribing COC.

ELIGIBILITY:
Inclusion Criteria:

* Women who had an episode of documented VTE (deep vein thrombosis and / or pulmonary embolism) under COC who consulted in a specialized counseling center.
* Women of age.
* Subject agreeing to participate in this research, having signed informed consent.

Exclusion Criteria:

* Absence of COC,
* No knowledge of the COC generation used by the patient,
* Undocumented MTEV Episode
* Absence of available sample (DNA),
* Refusal to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1454 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-09 (Actual)

PRIMARY OUTCOMES:
Build a predictive score for VTE in women using COC | 42 months
  this score is based on clinical and biological factors

CONTACTS AND LOCATIONS:
Overall Officials: jean-olivier ARNAUD, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France